CLINICAL TRIAL: NCT02309229
Title: Sputum Purulence as a Predictor of Cystic Fibrosis Exacerbations: a Prospective Cohort Trial.
Acronym: MucoSpuCo
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Lieven Dupont, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML8808; S54884 (Other: UZ Leuven)
Record Dates: First submitted 2013-04-05; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis
Keywords: sputum colour; cystic fibrosis; pollution
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cystic fibrosis patients: patients with cystic fibrosis

SUMMARY:
To use the sputum colour chart as a predictor for cystic fibrosis exaerbations

DETAILED DESCRIPTION:
Patients will score their sputum purulence daily using three colour charts. They will also score for respiratory and other symptoms.

Primary analysis will focus on the predicting value of sputum purulence on exacerbations. Secondary analysis will evaluate symptoms on exacerbation prediction. A third subanalysis will focus on correlation of daily pollution fluctuations and sputum purulence or symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of cystic fibrosis
* Pseudomonas aeruginosa colonization
* at least 2 exacerbations in the previous year
* at least 18 years of age

Exclusion Criteria:

* colour blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
sputum colour evoluation as a predictor for exacerbation | 6 months

SECONDARY OUTCOMES:
symptoms as a predictor for exacerbations | 6 months

OTHER OUTCOMES:
pollution and symptoms/exacerbations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lieven J Dupont, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University hospital Leuven, Leuven, Vlaams-Brabant, Belgium